CLINICAL TRIAL: NCT07373535
Title: Toward Patient-Tailored Care for Treatment-Resistant Depression: A Pilot Patient-Preference Clinical Trial of Music and Mindfulness in Psilocybin-Assisted Psychotherapy
Brief Title: Understanding Music and Mindfulness Preferences in Psilocybin-Assisted Psychotherapy
Acronym: PPP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyle Greenway (Other)
Responsible Party: Sponsor-Investigator, Kyle Greenway, Psychiatrist and Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-4333; 288527 (Other: Health Canada)
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Treatment-Resistant Major Depressive Disorder
Keywords: Psilocybin; Clinical Trial; Depressive Disorder, Treatment-Resistant; Music; Mindfulness; Feasibility; Culture; Patient preference
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Patient Preference | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: A 10-week, pilot patient-preference clinical trial with two four-week treatment phases.
  At baseline, enrolled patients with TRD will rate their preferences for music-centered and mindfulness-centered approaches to PAP.
  Treatment phase one (weeks 1-4): patients will receive either their preferred or non-preferred treatment approach over 4 weeks, based on a simple 50:50 randomization.
  The key endpoint will occur in week 5. No treatment will take place between weeks 5-6. Treatment phase two (weeks 7-10): patients will be crossed-over to receive the other treatment approach over four weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preferred treatment (Experimental)
  Interventions: Drug: Psilocybin 25mg; Other: Music-centered psilocybin-assisted therapy; Other: Mindfulness-centered psilocybin-assisted therapy
- Non-preferred treatment (Experimental)
  Interventions: Drug: Psilocybin 25mg; Other: Music-centered psilocybin-assisted therapy; Other: Mindfulness-centered psilocybin-assisted therapy

INTERVENTIONS:
Drug: Psilocybin 25mg — Psilocybin 25mg
  Other Names: PEX010(25)
Other: Music-centered psilocybin-assisted therapy — Psilocybin therapy emphasizing the use of music.
Other: Mindfulness-centered psilocybin-assisted therapy — Psilocybin therapy emphasizing the use of guided mindfulness.

SUMMARY:
The goal of this pilot clinical trial is to learn whether it is feasible to individually tailor psilocybin-assisted psychotherapy (PAP) for people with treatment-resistant depression (TRD) based on their personal preferences. The study also aims to explore whether two different psychotherapy styles, music-centered and mindfulness-centered, influence how people respond to psilocybin treatment.

The main questions it aims to answer are:

* Is it feasible to conduct a patient-preference randomized trial of psilocybin-assisted psychotherapy?
* Does receiving a preferred psychotherapy style improve treatment experiences or outcomes?
* How do music-centered and mindfulness-centered PAP approaches compare in their effects on improving mood and well-being?

Researchers will compare music-centered PAP to mindfulness-centered PAP to see if aligning psychotherapy with individual preferences is a practical and potentially beneficial approach for improving treatment efficacy and tolerability.

Participants will:

* Be adults with treatment-resistant depression
* Receive two 25 mg psilocybin (PEX010, Filament Health) sessions, spaced four weeks apart
* Experience one session with music-centered psychotherapy and one with mindfulness-centered psychotherapy
* Before treatment, rate their preference for the two psychotherapy approaches
* Be randomly assigned to receive their preferred or non-preferred approach first, followed by the other
* Complete preparation and integration sessions before and after each psilocybin session

This feasibility trial will also collect information on participants' cultural and personal factors influencing psychotherapy preferences using a modified Cultural Formulation Interview, and explore physiological measures of therapeutic alliance, an important factor in psychotherapy outcomes.

DETAILED DESCRIPTION:
Depression is one of the top causes of disability worldwide. Psilocybin-assisted psychotherapy (PAP) is an emerging treatment for Treatment-Resistant Depression (TRD) that pairs one or two doses of psilocybin, a serotonergic psychedelic, with a brief course of psychotherapy. While multiple studies of PAP have found safe, rapid, and lasting antidepressant effects, much remains unknown about how to optimize this promising intervention's psychotherapy component.

This pilot study aims to explore a novel strategy for improving the efficacy and tolerability of PAP: individually-tailoring its psychotherapy based on patient preferences for two important nonpharmacological treatment elements: music and mindfulness. These core treatment components were selected based on their ubiquitousness in psilocybin studies and their potential for significant patient preference effects.

The investigators will conduct a patient-preference randomized clinical trial where 16 patients with TRD will receive two doses of psilocybin (PEX010, Filament Health, 25mg). For each patient, one psilocybin dose will be administered with music-centered psychological support and the other with mindfulness-centered psychological support. In the first 4-week phase, patients will be asked to rate their preferences for these different psychotherapeutic approaches. Patients will then be 50:50 randomized to first receive either their preferred or their non-preferred treatment approach. In a second 4-week crossover phase, patients will receive the other treatment approach. All patients will thus undergo both music-centered and mindfulness-centered PAP interventions, but in an order dictated by their preferences and randomization. Each treatment phase entails pre-treatment and post-treatment psychotherapy following standard protocols.

Similar patient-preference clinical trial designs have shown that preferences can significantly influence the efficacy and tolerability of existing psychiatric treatments. The primary aim of this pilot trial is to examine this design's feasibility for exploring such preference effects in PAP, which the investigators hypothesize will be substantial. As secondary aims, the trial will generate preliminary estimates about the magnitude of preference effects, compare the music- and mindfulness-centered approaches, and yield qualitative data about the diverse sociocultural factors that influence patient preferences, including with a modified Cultural Formulation Interview administered at baseline. An additional exploratory aim is to examine novel physiological measures of therapeutic alliance, a crucial factor in psychiatric care.

Depression affects millions of Canadians and new treatments are sorely needed. This line of research seeks to produce systematic approaches to tailoring the psychotherapy of PAP for TRD. Its ultimate goal is to improve this promising intervention's efficacy, safety, and applicability to diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age at screening.
* Diagnosis of unipolar Major Depressive Disorder (MDD) according to diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5-TR), confirmed by a study psychiatrist using the Mini International Neuropsychiatric Interview (MINI) version 7.0.2.
* Failure to achieve remission from at least two trials of evidence-based oral antidepressants, in the current episode, of adequate dose and duration.
* Moderate to severe symptoms according to the clinician-administered Montgomery-Åsberg Depression Rating Scale (MADRS): total score ≥ 25 on screening.
* Active follow-up in psychiatry.
* Able and willing to give informed consent to participate in the study, and for the study clinicians to communicate with their psychiatrist throughout the intervention phase of the study.
* Available and willing to comply with all study assessments.
* Stable psychotropic medications for at least eight weeks at the time of enrollment.
* Able to read and understand French and/or English.
* Has at least one identified support person, including a friend or family member, who agrees to accompany patient home (or to an otherwise safe destination) following the psilocybin treatment sessions.

Exclusion Criteria:

* Deemed to be greater than low risk of suicide on psychiatric interview.
* Currently or previously diagnosed with any of the following, according to available information and psychiatric interview: major depression with psychotic features, schizophrenia spectrum or other psychotic disorders, and/or bipolar affective disorder I or related disorders.
* Current or past diagnosis of personality disorder deemed to pose a significant risk for safety and/or trial compliance.
* Family history (first-degree relative) of psychosis.
* Current or recent (< six months) substance use disorder, except for tobacco use disorder.
* Deemed to be greater than low risk of future substance use disorder.
* Currently receiving and deemed to be unsuitable, on psychiatric interview, to discontinue medications with significant serotonin 2A antagonism (e.g., trazodone) or known potential for serious interactions with psilocybin including serotonin syndrome (e.g., monoamine oxidase inhibitors), seizures (e.g., lithium), or which may affect psilocybin pharmacokinetics (e.g. UDG modulators, aldehyde dehydrogenase inhibitors).
* Unwilling or unable to maintain current psychotropic medications throughout the treatment phase of the trial.
* Currently undergoing psychotherapy that will not remain stable for the duration of the study or was initiated within 21 days of baseline.
* Prior use of serotonergic psychedelics in the past year and/or more than five life-time uses.
* Use of any serotonergic psychedelic or ketamine, or any other illicit substance during the active treatment period of the trial.
* Medical contraindications:
* Current or past history of seizure disorder with the exception of infantile febrile seizures.
* Significant cardiovascular disease including uncontrolled blood pressure (> 140/90mmHg), clinically significant arrhythmia, heart failure, coronary artery disease, history of ischemic or hemorrhagic stroke, or history of myocardial infarction.
* Abnormal and clinically significant results on the physical examination, laboratory investigations, or ECG at screening.
* Any other clinically significant illness deemed to pose significant health risks for participation in the study.
* Pregnant or lactating.
* For women of child-bearing potential, defined as all women physiologically capable of becoming pregnant: unwilling to utilize highly effective contraceptive during the 10-week active intervention (e.g., oral contraceptive). Acceptable forms of highly effective contraception methods include: a. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception; b. Male/female sterilization defined as: 1) Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed and documented by follow up hormone level assessment; 2) Male sterilization of the sole partner (at least 6 months prior to screening) of a female patient on the study. c. A combination of any two of the following (i+ii or i+iii or ii+iii):

  i) Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository ii) Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception iii) Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Men unwilling to not attempt to father a child or not donate sperm, while participating the active treatment period of this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Enrollment Feasibility | From screening through enrollment
  The proportion of participants screened as eligible who enroll in the trial.
Overall Trial Completion Feasibility | From enrollment through the end of active treatment (Week 10)
  The proportion of enrolled participants who complete the trial, defined as attending ≥ 90% of required study visits.
Trial Completion by Preference Assignment | From enrollment through the end of active treatment (Week 10)
  The proportion of participants in the preferred and non-preferred treatment groups who complete ≥ 90% of study visits.
Distribution of Treatment Preferences | Baseline
  The proportion of participants who choose the music-centered versus the mindfulness-centered approach as their preferred treatment at baseline.
Ease of Delivering Treatment Approaches as Assessed by the NASA-TLX | End of each psilocybin treatment session (Week 3, Week 9)
  The ease of delivering the music-centered versus the mindfulness-centered as assessed by therapists' reported levels of effort with each intervention measured with the NASA Task Load Index (NASA-TLX). The NASA Task Load Index (NASA-TLX) is a self-reported measure assessing perceived workload and cognitive effort during a task that will be completed by the therapists. It evaluates six dimensions: Mental Demand, Physical Demand, Temporal Demand, Performance, Effort, and Frustration. Each dimension is rated using a continuous 0-100 visual analog scale, with anchors ranging from very low (0) to very high (100) (for Performance, 0 = poor to 100 = excellent). Higher scores reflect greater perceived workload, except for Performance, where higher scores indicate better perceived performance. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered vs. mindfulness-centered).
Theoretical Framework of Acceptability (TFA) | Baseline, Weeks 3 and 9 (treatment sessions), Week 11 (follow-up)
  Acceptability of each therapeutic approach as measured by the Theoretical Framework of Acceptability (TFA) questionnaire for music-centered and mindfulness-centered interventions.
  Items cover comfort with the intervention, effort required, ethical or moral concerns, perceived effectiveness, clarity of intervention rationale, confidence in performing required activities, potential interference with other priorities, and overall acceptability. Each item is rated on a 5-point Likert scale (1 = lowest to 5 = highest). Total scores are calculated by summing all item responses, with possible scores ranging from 8 to 40. Higher scores indicate greater acceptability of the intervention.

SECONDARY OUTCOMES:
Rate of Adverse Events in Music- versus Mindfulness-centered Interventions | Baseline, Week 5 (primary endpoint), Week 11 (follow-up)
  Rates of adverse events in participants receiving music-centered versus mindfulness-centered approaches. Adverse events include any treatment-emergent symptoms reported by participants or observed by study staff.
Rate of Adverse Events in Preferred vs. Non-Preferred Interventions | Baseline, Week 5 (primary endpoint), Week 11 (follow-up)
  Rates of adverse events in participants receiving their preferred versus non-preferred interventions. Adverse events include any treatment-emergent symptoms reported by participants or observed by study staff.
Rate of Participant Drop-Outs in Preferred vs. Non-Preferred Interventions | Baseline, Week 5 (primary endpoint), Week 11 (follow-up)
  Rates of participant drop-outs in participants receiving their preferred versus non-preferred interventions. Drop-out is defined as missing more than 10% of scheduled visits during the active treatment period.
Rate of Participant Drop-Outs in Music- versus Mindfulness-centered Interventions | Baseline, Week 5 (primary endpoint), Week 11 (follow-up)
  Rates of participant drop-outs in participants receiving music-centered versus mindfulness-centered approaches. Drop-out is defined as missing more than 10% of scheduled visits during the active treatment period.
Change From Baseline in MADRS Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Montgomery-Åsberg Depression Rating Scale is a 10-item, clinician-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 6 (item's symptoms are severe). The total possible score is 60. Higher scores indicate greater severity. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in BDI-II Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Beck Depression Inventory Scale is a 21-item, patient-rated scale to rate the severity of the depressive symptoms. Each item is scored from 0 (item's symptoms not present) to 3 (item's symptoms are severe). The total possible score is 63. Higher scores indicate greater severity. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in GAD-7 Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item, participant-rated measure assessing the core symptoms of generalized anxiety over the past two weeks. Each item is scored from 0 (not at all) to 3 (nearly every day), yielding a total score from 0 to 21. Higher scores indicate greater severity of anxiety symptoms. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in the 5-level EQ-5D version (EQ-5D-5L) Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The EQ-5D-5L is a standardized, self-reported measure of health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-level scale reflecting increasing severity of problems. Responses are converted into a single index score, ranging from -0.59 to 1, with 1 representing the best possible health state. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) is a self-reported measure of enjoyment and satisfaction across multiple domains of daily functioning, including physical health, mood, work, household activities, social relationships, and general activities. The total score is calculated as the sum of the first 14 items, each rated on a 5-point Likert scale ranging from 1 (very poor) to 5 (very good). Total scores range from 14 to 70, with higher scores indicating greater enjoyment and satisfaction with quality of life. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in Work and Social Adjustment Scale (WSAS) Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Work and Social Adjustment Scale (WSAS) is a 5-item, self-reported measure of functional impairment attributable to a mental health problem across five domains: work, home management, social leisure activities, private leisure activities, and close relationships. Each item is rated on a 9-point scale ranging from 0 (no impairment) to 8 (severe impairment). Total scores range from 0 to 40, with higher scores indicating greater functional impairment. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in Gratitude Questionnaire-Six Item Form (GQ-6) Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Gratitude Questionnaire-Six Item Form (GQ-6) is a 6-item, self-reported measure of dispositional gratitude. Items are rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Total scores are calculated by summing item responses, with possible scores ranging from 6 to 42. Higher scores indicate greater levels of gratitude. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in Multidimensional Psychological Flexibility Inventory (MPFI-24) Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Multidimensional Psychological Flexibility Inventory-24 item version (MPFI-24) is a self-reported measure of psychological flexibility across six core processes: acceptance, defusion, present-moment awareness, self-as-context, values, and committed action. Items are rated on a 6-point Likert scale ranging from 1 (never true) to 6 (always true). The total score is calculated by summing item responses after appropriate reverse scoring of psychological inflexibility items. Total scores range from 24 to 144, with higher scores indicating greater psychological flexibility. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in Watts Connectedness Scale (WCS) Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Watts Connectedness Scale (WCS) is a self-reported measure of perceived psychological and existential connectedness, including connectedness to self, others, nature, and the broader universe. The scale consists of 23 items rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Total scores are calculated by summing item responses, with possible scores ranging from 23 to 161. Higher scores indicate greater perceived connectedness. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Change From Baseline in Pearlin Mastery Scale Total Score to Key Endpoint | Baseline, Week 5 (primary endpoint)
  The Pearlin Mastery Scale is a 7-item, self-reported measure of perceived control over life circumstances. Items are rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). Total scores are calculated by summing item responses, with possible scores ranging from 7 to 28. Higher scores indicate a greater sense of mastery or perceived control. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Semi-structured Qualitative Interviews | Baseline, Week 11 (follow-up)
  The Cultural Formulation Interview, adapted for psychedelic therapy, will be used identify of factors relevant to participants' experiences and preferences at baseline. Post-trial interviews will be conducted to capture factors that influence the participants' experiences and treatment preferences.
Challenging Experience Questionnaire Brief (CEQ-7) | End of each psilocybin treatment session (Week 3, Week 9)
  The Challenging Experience Questionnaire-7 item version (CEQ-7) is a self-reported measure assessing the intensity of challenging experiences during a treatment session. Participants rate 7 statements on a 6-point Likert scale ranging from 0 (not at all) to 5 (extremely). Total scores are calculated by summing all item responses, with possible scores ranging from 0 to 35. Higher scores indicate greater intensity of challenging experiences. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Acceptance/Avoidance-Promoting Experiences Questionnaire (APEQ-SF) | End of each psilocybin treatment session (Week 3, Week 9)
  The Acceptance/Avoidance-Promoting Experiences Questionnaire - Short Form (APEQ-SF) is a 21-item, self-reported measure assessing the extent to which participants experience acceptance-promoting versus avoidance-promoting psychological processes during a treatment session. Items are answered dichotomously as 0 (No, not at all) or 1 (Yes, extremely or absolutely). Total scores are calculated by summing item responses, with possible scores ranging from 0 to 21. Higher scores indicate greater engagement in acceptance-promoting experiences relative to avoidance. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Imprinting (Self-constructed) | End of each psilocybin treatment session (Week 3, Week 9)
  The Imprinting Questionnaire is a 5-item, self-reported measure assessing the extent to which participants experience hallucinations influenced by previously seen content. Items include vivid visual hallucinations, hallucinations resembling recently or previously seen media (e.g., television, video games, paintings), and hallucinations resembling recently or previously seen non-media scenes (e.g., landscapes, cities). Participants respond dichotomously (0 = No, not at all; 1 = Yes, extremely or absolutely). Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Mystical Experience Questionnaire Brief (MEQ-4) | End of each psilocybin treatment session (Week 3, Week 9)
  The Mystical Experience Questionnaire-4 item version (MEQ-4) is a self-reported measure assessing the intensity of mystical-type experiences during a treatment session. Participants rate 4 statements on a 6-point Likert scale ranging from 0 (none) to 5 (extreme). Total scores are calculated by summing all item responses, with possible scores ranging from 0 to 20. Higher scores indicate stronger mystical-type experiences. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Awe Experience Scale - Short Form (AWE-SF) | End of each psilocybin treatment session (Week 3, Week 9)
  The Awe Experience Scale - Short Form (AWE-SF) is a 12-item, self-reported measure assessing the intensity of awe experienced during a treatment session across six factors: Time, Self-Loss, Connectedness, Vastness, Physiological Changes, and Accommodation. Items are rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Total scores are calculated by averaging all item responses, with possible scores ranging from 1 to 7. Higher scores indicate stronger experiences of awe. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Modified Psychedelic Communitas Scale | End of each psilocybin treatment session (Week 3, Week 9)
  The Modified Psychedelic Communitas Scale is an 8-item, self-reported measure assessing the sense of relational connection, shared humanity, and social bonding experienced with facilitators during a treatment session. Items include feeling a bond, a sense of belonging, harmony, sharing, equality, irrelevance of social status, resolution of ego-related tensions, and strong connection with facilitators. Participants rate each item on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Total scores are calculated by summing item responses, with possible scores ranging from 8 to 56. Higher scores indicate stronger communitas experiences. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Psychedelic Music Questionnaire Short-Form (PMQ-SF) | End of each psilocybin treatment session (Week 3, Week 9)
  The Psychedelic Music Questionnaire - Short Form (PMQ-SF) is a self-reported measure assessing participants' experiences of music during a psychedelic treatment session. Items assess the extent to which the music was supportive, meaningful, personally resonant, aesthetically appreciated, emotionally engaging, and helped participants gain new insights, as well as any negative reactions such as feeling distracted, irritated, or unsafe. Participants rate 15 items on a 5-point Likert scale ranging from 1 (not at all) to 5 (extremely). Total scores are calculated by summing item responses, with possible scores ranging from 15 to 75. Higher scores indicate more positive and engaging experiences with the music. Scores will be compared by preference group (preferred vs. non-preferred) .

OTHER OUTCOMES:
Therapeutic Alliance - Patient (WAI-SR) | Weeks 1 and 7 (preparation sessions), Weeks 3 and 9 (treatment and integration sessions)
  The Working Alliance Inventory - Short Revised (WAI-SR, Patient version) is a 12-item, self-reported measure assessing patients' perception of the therapeutic alliance during treatment sessions. Items assess agreement, collaboration, and bond with the therapist, including understanding goals, agreement on tasks, mutual respect, and perceived care and support. Participants rate each item on a 5-point Likert scale ranging from 1 (seldom) to 5 (always). Total scores are calculated by summing item responses, with possible scores ranging from 12 to 60. Higher scores indicate a stronger therapeutic alliance. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Therapeutic Alliance - Therapist (WAI-SRT) | Weeks 1 and 7 (preparation sessions), Weeks 3 and 9 (treatment and integration sessions)
  The Working Alliance Inventory - Short Revised (WAI-SR, Therapist version) is a 10-item, self-reported measure assessing therapists' perception of the therapeutic alliance during treatment sessions. Items evaluate agreement on goals and tasks, mutual understanding, collaboration, respect, and concern for the patient's welfare. Therapists rate each item on a 5-point Likert scale ranging from 1 (seldom) to 5 (always). Total scores are calculated by summing item responses, with possible scores ranging from 10 to 50. Higher scores indicate a stronger perceived therapeutic alliance. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Linguistic Synchrony | Weeks 1 and 7 (preparation sessions), Weeks 3 and 9 (treatment and integration sessions)
  Linguistic synchrony between the participant and clinicians will be quantified using Natural Language Processing (NLP) applied to session transcripts. The measure has no predefined minimum or maximum value; higher values indicate greater alignment in language use between the participant and clinicians. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).
Cardiovascular Synchrony | Weeks 1 and 7 (preparation sessions), Weeks 3 and 9 (treatment and integration sessions)
  Cardiovascular synchrony between the participant and clinicians will be assessed using electrocardiography (ECG)-derived heart rate variability (HRV) and respiratory sinus arrhythmia (RSA). A validated surrogate synchrony method will be applied to quantify the extent of physiological alignment between the participant and clinicians during therapy sessions. The measure has no predefined minimum or maximum value; higher values indicate greater cardiovascular synchrony. Scores will be compared by preference group (preferred vs. non-preferred) and therapeutic approaches (music-centered versus mindfulness-centered).

CONTACTS AND LOCATIONS:
Overall Officials: Kyle T Greenway, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No